CLINICAL TRIAL: NCT00938210
Title: Changes in Fatigue and Physical Function Following Laparoscopic Colonic Surgery
Brief Title: Rehabilitation Following Laparoscopic Colonic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Martin Bach Jensen, Associate Professor, Institute of Public Health Aarhus, Aarhus University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBJ-1
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Colonic Cancer; Postoperative Care; Fatigue
Keywords: Colonic surgery; Postoperative care; Fatigue; Physical function; Quality of life
MeSH Terms: conditions — Colonic Neoplasms; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Laparoscopic surgery (No Intervention): Patients undergoing laparoscopic colonic surgery are compared with a historical cohort of patients undergoing similar open colonic surgery (right hemicolectomy and sigmoid resections).
  Interventions: Procedure: Laparoscopic colonic surgery

INTERVENTIONS:
Procedure: Laparoscopic colonic surgery — Laparoscopic removal of colonic cancer

SUMMARY:
The standard procedure for treating colonic cancer is changing from open surgery to laparoscopic surgery. Following open colonic surgery patients are fatigued and loss body mass and have a reduction in physical function, but the investigators do not know if this is also the case following laparoscopic surgery.

This study examines how fatigue, quality of life, physical function, and body composition changes following laparoscopic colonic surgery.

Patients are examined preoperatively and postoperative day 10 and 30.

ELIGIBILITY:
Inclusion Criteria:

* elective colonic cancer surgery
* hemicolectomy or sigmoid resection
* informed consent

Exclusion Criteria:

* disseminated cancer
* contraindications for laparoscopic surgery
* dementia or serious psychiatric disease
* diseases or other aspects that prohibit participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-05; Primary Completion 2011-11 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Fatigue | Preoperative to postoperative day 10

SECONDARY OUTCOMES:
Muscular strength | From preoperatively to postoperative day 10 and 30
Change in work capacity (pulse rate) | From pre- to postoperative day 10 and 30
Balance (sway) | From preoperatively to postoperative day 10 and 30
Pain at rest and when moving | From preoperatively to postoperative day 10 and 30
Quality of life (Short Form 36 - SF-36) | From preoperatively to postoperative day 10 and 30
Body weight | From preoperatively to postoperative day 30
Body composition (fat mass and fat free mass estimated by bio-impedance) | From preoperatively to postoperative day 10 and 30
Social support | From preoperatively to postoperative day 10 and 30

CONTACTS AND LOCATIONS:
Overall Officials: Martin B Jensen, MD, Ph.d., Principal Investigator — Research Unit for General Practice in the North Denmark Region, Institute of Public Health, Aarhus University; Søren Laurberg, Professor, Study Chair — Department of Surgery P, Aarhus University Hosptial
Locations (2):
- Denmark (2):
  - Department of Surgery, Herning Hospital, Herning
  - Department of Surgery, Randers